CLINICAL TRIAL: NCT01984060
Title: Feasibility of an Exercise Intervention In HIV+ Older Adults
Brief Title: Feasibility of an Exercise Intervention
Acronym: MESH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Krupa Shah, M.D. Assistant professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1K23AG043319-01A1 (NIH)
Record Dates: First submitted 2013-10-24; First posted 2013-11-14 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: HIV
Keywords: Aging; Physical Activity; Physical Function; HIV; Frailty; Autonomous Motivation; Depression
MeSH Terms: conditions — Motor Activity; Frailty; Depression

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- HOME-EX (Other): Motivational Counseling: Six patient-centered motivational counseling sessions based on the self-determination theory (SDT) of behavior change will be conducted with the patients in the HOME-EX group over 12 weeks.
  Exercise Intervention: an individually tailored home-based exercise program performed 5-7 days a week that consists of walking prescription, and individualized strength training exercise designed to provide moderately intense progressive resistance exercise. Subjects will be given a set of 3 color-coded therapeutic resistance bands representing varying levels of resistance and they will start with a number of sets which is customized for each individual and they will be encouraged to progressively increase from their individual baseline sets.
  Interventions: Other: HOME-EX
- Control (No Intervention): Subjects are instructed to maintain their usual activities during the study period. This group did not receive any PA counseling or recommendations.

INTERVENTIONS:
Other: HOME-EX — Motivational Counseling: The first session will be an hour face-to-face interview to establish a rapport with subjects, assess motives and competence. The rest will be 30 min. phone calls to assess week's performance and agree on an action plan for next 2 weeks.
  Exercise Intervention: Using the average number of steps for each subject from their baseline assessment, the targeted number of steps the subject needs to walk every day will be calculated. The individualized strength training exercise will target the upper and lower body. If possible, they will be encouraged to progressively increase from their individual baseline sets and repetitions to a maximum of 4 sets of 15 repetitions for each exercise
  Arms: HOME-EX

SUMMARY:
The overall purpose of this research is to evaluate the effect of a home-based exercise program on physical function and to improve the health and quality of life for the HIV-infected older adult community.

DETAILED DESCRIPTION:
Subjects are being asked to participate in this study if they are infected with the human immunodeficiency virus (HIV), and they are 45 years of age or older.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive, both genders, all races, English speaking individuals, age 45 years or older, on HAART before enrollment. .

Exclusion Criteria:

* Subject will be excluded if he/she has history or currently has severe cardiopulmonary illness, severe orthopedic or neuromuscular impairments, significant cognitive or sensory impairments, history of active malignancy, untreated depression, manic or psychotic disorder, and normal PPT score.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-12; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in Feasibility | At day zero of the study and after 12 weeks of intervension.
  To develop and establish the feasibility of home-exercise(HOME-EX)in HIV positive subjects as evaluated by measuring exercise adherence and acceptability, exercise intensity and adverse events. We hypothesize that HOME-EX is a feasible and safe intervention for HOA.

SECONDARY OUTCOMES:
Change in Efficacy | At day zero of the study and after 12 weeks of intervension.
  To determine the potential efficacy of HOME-EX in HIV positive adults in improving physical function as evaluated by the physical performance test (PPT). We hypothesize that physical function will improve in the HOME-EX group compared to the CONTROL group.
Change in Autonomy | At day zero of the study and after 12 weeks of intervension.
  To determine the potential efficacy of HOME-EX in HIV positive on exercise-related psychological mediators as evaluated by the SDT-based questionnaires. We hypothesize that the HOME-EX group will report greater perceived autonomy support, more autonomous self-regulation, higher intrinsic motivation and perceived competence compared to the CONTROL group.

CONTACTS AND LOCATIONS:
Overall Officials: Krupa Shah, M.D., M.P.H., Principal Investigator — University of Rochester
Locations (1):
- University of Rochester/ Strong Memorial Hospital, Rochester, New York, United States

REFERENCES:
- [Derived] Shah KN, Majeed Z, Yoruk YB, Yang H, Hilton TN, McMahon JM, Hall WJ, Walck D, Luque AE, Ryan RM. Enhancing physical function in HIV-infected older adults: A randomized controlled clinical trial. Health Psychol. 2016 Jun;35(6):563-73. doi: 10.1037/hea0000311. Epub 2016 Feb 11. PMID 26867045